CLINICAL TRIAL: NCT06831656
Title: The Effect of TetraSOD® Supplementation on Blood Oxidative Stress Biomarkers and Endurance Exercise Performance in Healthy Adults
Brief Title: TetraSOD® Supplementation and Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Fitoplancton Marino, S.L. (Industry)
Responsible Party: Principal Investigator, Stephen Bailey, Reader in Human and Exercise Physiology, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R19-P160
Record Dates: First submitted 2024-12-31; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-12

CONDITIONS: Placebo-Pre; Placebo-Post; Tetraselmis Chuii-Pre; Tetraselmis Chuii-Post
Keywords: Microalgae; Endurance performance

STUDY DESIGN:
Intervention Model Description: Crossover Assignment 13 participants completed 2 experimental conditions in a randomized order.
Who Masked: Participant, Investigator
Masking Description: Funder
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo-Pre (Other): No supplementation prior to undergoing the placebo supplement
  Interventions: Other: Placebo-Pre
- Placebo-post (Placebo Comparator): Placebo supplementation
  Interventions: Dietary Supplement: Placebo-Post
- Tetraselmis chuii-Pre (Other): No supplementation prior to undergoing the Tetraselmis chuii supplement
  Interventions: Other: Tetraselmis chuii-Pre
- Tetraselmis chuii-Post (Active Comparator): Tetraselmis chuii supplementation
  Interventions: Dietary Supplement: Tetraselmis chuii-Post

INTERVENTIONS:
Other: Placebo-Pre — No dietary supplementation prior to undergoing the placebo supplement
  Arms: Placebo-Pre
Dietary Supplement: Placebo-Post — 14 days of supplementation with 25 mg/day hemicellulose crystalline
  Arms: Placebo-post
Other: Tetraselmis chuii-Pre — No dietary supplementation prior to undergoing the tetraselmis chuii supplement
  Arms: Tetraselmis chuii-Pre
Dietary Supplement: Tetraselmis chuii-Post — 14 days of supplementation with 25 mg/day tetraselmis chuii
  Arms: Tetraselmis chuii-Post

SUMMARY:
Tetraselmis chuii (TetraSOD) is a marine microalgae that has been reported to improve antioxidant responses in human skeletal muscle cells treated with TetraSOD and to improve recovery from muscle damaging exercise in humans supplemented with TetraSOD. However, the effects of TetraSOD supplementation on endurance performance and physiology is less clear. This study assessed the effect of short-term TetraSOD supplementation on endurance performance and physiology in healthy adults.

DETAILED DESCRIPTION:
It is well documented that the production of reactive oxygen species (ROS; unstable molecules that react easily with and damage other molecules in a cell) increases in-line with the intensity and duration of exercise . Although increased ROS production during exercise is initially managed by a variety of 'antioxidants', continued ROS production exceeds the capacity of this antioxidant defense system leading to the development of oxidative stress and impaired exercise performance. Therefore, interventions that can lessen exercise-induced oxidative stress have the potential to improve exercise performance. While dietary supplementation with antioxidant vitamins (e.g. vitamin C and E) has this potential, such interventions do not typically improve exercise performance.

Therefore, further research is required to investigate the potential for novel nutritional supplements to lessen exercise-induced oxidative stress and to improve exercise performance.

Tetraselmis chuii (TetraSOD) is a natural marine microalgae product. Recent preliminary evidence suggests that treating human skeletal muscle cells with TetraSOD can increase the production of antioxidant enzymes to limit oxidative stress development. In addition, TetraSOD supplementation has been reported to improve recovery from muscle damaging exercise. However, the effects of TetraSOD supplementation on endurance performance and physiology is less clear.

The purpose of this study was to assess the effect of short-term TetraSOD supplementation on endurance performance and physiology in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male (as determined by the Health Screening Questionnaire)
* Adult (aged ≥18 and ≤40 years old)
* Recreationally-active (≥2 and ≤4 exercise sessions per week) and a V̇O2max of ≥ 35 mL/kg/min and ≤ 65 mL/kg/min as determined from the preliminary exercise test
* No known history of gastric, digestive, cardiovascular, renal disease or any other orthopaedic diseases related to motor organs
* Non-smoker
* Healthy body mass index (BMI; ≥18.5 and ≤24.9 kg/m2)
* Not using any dietary supplements, including antioxidant and nitrate-rich supplements, currently or in the past one month
* Not a heavy drinker (≤ 14 units of alcohol) on most weeks
* Not using medication that may affect study measures
* Not participating in other studies currently or in the past two months prior to the consenting session (visit 1) or having an intention to participate in other studies over the period of this study

Exclusion Criteria:

* Female
* Aged <18 and >40 years old
* Sedentary or highly trained with a respective V̇O2max of < 35 mL/kg/min and > 65 mL/kg/min as determined from the preliminary exercise test
* History of gastric, digestive, cardiovascular, renal disease or any other orthopaedic diseases related to motor organs
* Smoker
* Unhealthy body mass index (BMI;<18.5 and >24.9 kg/m2)
* Using any dietary supplements, including antioxidant and nitrate-rich supplements, currently or in the past one month
* Heavy drinker (> 14 units of alcohol) on most weeks
* Using medication that may affect study measures
* Participating in other studies currently or in the past two months prior to the consenting session (visit 1) or having an intention to participate in other studies over the period of this study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion during a severe-intensity cycle ergometry test continued until exhaustion | One assessment prior to and 14 days following the placebo supplementation, and one assessment prior to and 14 days following Tetraselmis chuii supplementation
  Time to exhaustion during severe-intensity cycle ergometry measured in seconds
End-exercise pulmonary oxygen uptake during a severe-intensity cycle ergometry test continued until exhaustion measured using an online gas analyser | One assessment prior to and 14 days following the placebo supplementation, and one assessment prior to and 14 days following Tetraselmis chuii supplementation
  Pulmonary oxygen uptake at the end of a severe-intensity cycling bout completed until exhaustion to provide an estimate of VO2max measured in L/min using a breath-by-breath gas exchange analyzer and taken as the mean over the final 30 s of the test.

SECONDARY OUTCOMES:
End-exercise blood lactate concentration during a severe-intensity cycle ergometry test continued until exhaustion | One assessment prior to and 14 days following the placebo supplementation, and one assessment prior to and 14 days following Tetraselmis chuii supplementation
  Blood lactate concentration at the end of a severe-intensity cycling bout continued until exhaustion measured in mmol/L using an autoanalyzer
End-exercise rating of perceived exertion using the Borg 6-20 scale during a severe-intensity cycle ergometry test continued until exhaustion | One assessment prior to and 14 days following the placebo supplementation, and one assessment prior to and 14 days following Tetraselmis chuii supplementation
  Assessment of rating of perceived exertion at the end of a severe-intensity cycling bout completed until exhaustion using the Borg 6-20 scale where 6 = no exercise and 20 = maximal exertion with measurement units of arbitrary units.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bailey, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom